CLINICAL TRIAL: NCT03790176
Title: Plasma, ELF and Intraperitoneal Pharmacokinetics of Ceftazidime/Avibactam in Critically Ill and Peritoneal Dialysis Patients
Brief Title: ZAVI APD ELF Protocol v2.2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Markus Zeitlinger (Other)
Responsible Party: Sponsor-Investigator, Markus Zeitlinger, Assoc. Prof. Priv. Doz. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Version 2.2 April 19, 2018
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Peritonitis; Pneumonia
MeSH Terms: conditions — Peritonitis; Pneumonia | interventions — Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: group A - patients on automated peritoneal dialysis group B - critically ill patients with pneumonia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - patients on automated peritoneal dialysis (Other): each of n=8 patients will receive one single intravenous infusion of ceftazidime/avibactam (CAZ/AVI) 2g/0.5g over two hours. Subsequently, PK of CAZ/AVI will be determined in plasma and peritoneal dialysis fluid (and urine, if applicable) at protocol-defined time points over 24 hours.
  Interventions: Drug: Intravenous Infusion
- B - critically ill patients with pneumonia (Other): following one intravenous dose of 2g/0.5g CAZ/AVI (which patients will receive based on clinical indication by their treating physician), PK of CAZ/AVI will be determined at protocol-defined time points over one dosing interval in plasma and in epithelial lining fluid (ELF).
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: Intravenous Infusion — see arm/group description. NO INTERVENTION IN STUDY GROUP B! PATIENTS OF GROUP B WILL RECEIVE CAZ/AVI INDEPENDENTLY FROM STUDY PARTICIPATION BASED ON DECISION OF THEIR TREATING PHYSICIAN

SUMMARY:
CAZ/AVI is a new antibiotic drug that is meant to be used for various indications including cIAI and nosocomial pneumonia. To date, limited data exists on PK of CAZ/AVI in patients undergoing peritoneal dialysis as well as on penetration of CAZ/AVI in ELF of critically ill patients. The present study is carried out to determine target site PK of CAZ/AVI in these two populations, in order to contribute to a more complete understanding of the drug's penetration to its site of action.

DETAILED DESCRIPTION:
Ceftazidime/Avibactam (CAZ/AVI) is a novel antibiotic drug that has recently become available. It consists of a β-lactam/β-lactamase fixed drug combination with an almost exclusively Gram-negative spectrum and is indicated for the treatment of:

* complicated intra-abdominal infections (cIAI)
* complicated urinary tract infection (cUTI), including pyelonephritis
* hospital-acquired pneumonia including ventilator-associated pneumonia (VAP)
* infections due to aerobic Gram-negative organisms in patients with limited treatment options.

It is common knowledge that in anti-infective therapy, sufficient drug delivery to the target site is essential for antimicrobial efficacy and prevention of bacterial resistance. Based on this premise, the present exploratory trial will focus on the pharmacokinetics (PK) of CAZ/AVI in two patient populations:

PART A will investigate PK of CAZ/AVI in plasma and peritoneal dialysis fluid of patients undergoing automated peritoneal dialysis (APD). After a single intravenous dose of the drug PK sampling of CAZ/AVI will be performed in plasma and in peritoneal dialysis fluid, respectively. On the one hand, this will help to assess intraperitoneal exposure to CAZ/AVI after intravenous administration. This information might be of crucial importance for patients with infections localized in the peritoneal space. On the other hand, this study will show whether and to which extent CAZ/AVI is cleared from the bloodstream after intravenous administration in patients undergoing APD and receiving CAZ/AVI as treatment of other systemic infections, e.g. nosocomial pneumonia. Both aspects will improve current information on CAZ/AVI PK in peritoneal dialysis.

PART B will determine steady-state plasma and epithelial lining fluid (ELF) concentrations of CAZ/AVI in critically ill patients receiving the drug for treatment of nosocomial pneumonia (including VAP) at the discretion of their treating physicians. Penetration of CAZ/AVI into ELF has already been assessed in healthy volunteers and amounted roughly to 30% of plasma exposure. However, several physiological factors determining the amount of drug eventually recovered in ELF might be altered in critical illness (hemodynamics, binding to plasma and/or tissue proteins, local inflammation processes etc). Thus, PK of CAZ/AVI in lungs of critically ill patients might significantly differ from healthy volunteers, and deriving ELF exposure solely from plasma pharmacokinetics might not be entirely reliable in this circumstance. Still, considering the premise mentioned above, this issue is of crucial importance. The present study will help to assess whether CAZ/AVI reaches its target site (for the indication of nosocomial pneumonia) in critically ill patients to a sufficient degree.

Taken together, the information retrieved by this study will contribute to a better understanding of CAZ/AVI's disposition in target compartments of two patient populations and corroborate (or challenge) current dosing recommendations.

ELIGIBILITY:
Inclusion criteria (PART A - PATIENTS UNDERGOING APD):

* Males or females aged between 18 and 85 years undergoing automated peritoneal dialysis (APD)
* Written informed consent given after being provided detailed information about the nature, risks, and scope of the clinical study as well as the expected desirable and adverse effects of the drug
* No legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study

Exclusion criteria (PART A - PATIENTS UNDERGOING APD):

* Known allergy or hypersensitivity against study drug or other beta-lactam antibiotics
* History of severe allergic or anaphylactic reactions to any medication
* Any systemic infection
* Peritonitis or catheter-related infection which required antibiotic treatment within 2 months prior to the start of the study
* Pregancy or, in case of women of child-bearing potential, lack of willingness to apply adequate contraception measures during study period
* Haemoglobin below 9 g/dl
* Other objections to participate in the study in the opinion of the investigator

Inclusion criteria (PART B - CRITICALLY ILL PATIENTS):

* Age above 18 years
* Intubated patients admitted to an intensive care unit of the Vienna general hospital (AKH) participating in this study
* Sequential organ failure assessment (SOFA) score > 6 at study inclusion
* Clinical diagnosis of nosocomial pneumonia or VAP
* Body mass index (calculated from measured or estimated body weight and height) between 18 and 40
* Therapy with CAZ/AVI at a dosage of 2g/0.5g three times daily (indication at the discretion of the treating physicians)

Exclusion criteria (PART B - CRITICALLY ILL PATIENTS):

* Known allergy or hypersensitivity against study drug or other beta-lactam antibiotics
* Any disease considered relevant for proper performance of the study, or risks to the patient, at the discretion of the investigator
* Impaired renal function denoted by an estimated GFR of <50 mL/min according to Cockroft-Gault at study inclusion
* Requiring hemofiltration or hemodialysis
* Pregnancy
* Other factors that preclude study participation in the opinion of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve (AUC) from 0 to 8 hours (AUC0-8) | on study days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No